CLINICAL TRIAL: NCT04312698
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase III Trial to Evaluate the Efficacy and Safety of D013, D326 and D337 Combination Therapy in Dyslipidemia Patients With Hypertension
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-386
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A83_03DL/HT1903
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Dyslipidemia Patients With Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental)
  Interventions: Drug: D013, D326, D337
- Comparator Group 1 (Placebo Comparator)
  Interventions: Drug: placebo of D013, D326, D337
- Comparator Group 2 (Placebo Comparator)
  Interventions: Drug: D013, placebo of D326, placebo of D337

INTERVENTIONS:
Drug: D013, D326, D337 — Experimental: Group 1 Patients assigned to this group are treated with D013, D326, D337
  Other Names: Drugs are consist of antihypertensive agent and antihyperlipidemic agent
  Arms: Experimental Group 1
Drug: placebo of D013, D326, D337 — Placebo Comparator: Group 1 Patients assigned to this group are treated with D326, D337, placebo of D013
  Other Names: Drugs are consist of antihypertensive agent and antihyperlipidemic agent
  Arms: Comparator Group 1
Drug: D013, placebo of D326, placebo of D337 — Placebo Comparator: Group 2 Patients assigned to this group are treated with D013, placebo of D326, placebo of D337
  Other Names: Drugs are consist of antihypertensive agent and antihyperlipidemic agent
  Arms: Comparator Group 2

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of CKD-386

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are diagnosed with Dyslipidemia Patients with Hypertension or are being administered anti-hypertension and anti-hypertension drugs after diagnosis.
2. Subjects who agreed to participate in this clinical trial voluntarily.

Exclusion Criteria:

1. Subjects who were satisfied specific blood pressure levels that measured at screening period.
2. Subjects who were satisfied specific lipid levels that measured at screening period.
3. Subjects who cannot participate in a clinical trial based on the PI's judgment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Change rate from baseline in LDL-C | 8 weeks after drug administrations
  Compare experimental group 1 with comparator group 1
Change from baseline in MSSBP | 8 weeks after drug administrations
  Compare experimental group 1 with comparator group 2

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Medical Center Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No